CLINICAL TRIAL: NCT00937781
Title: Molecular Prognostic Factor Analysis in Melanoma
Brief Title: Study of Tumor Tissue From Patients With Melanoma Treated on Clinical Trial EST-1690
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000631851; ECOG-E1690T1
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Gene Expression Profiling; Microarray Analysis; Polymerase Chain Reaction; Immunohistochemistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: RNA analysis
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: polymerase chain reaction
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at tumor tissue samples from patients with melanoma treated on clinical trial EST-1690.

DETAILED DESCRIPTION:
OBJECTIVES:

* To validate the prognostic role of several biomarkers suggested by gene expression profiling and tissue microarray (TMA) studies (e.g., NCOA3, SPP1, and RGS1) on the outcome associated with melanoma in the EST-1690 cohort using IHC analysis.
* To examine the potential predictive role of such biomarkers in patients undergoing adjuvant interferon alfa therapy.
* To analyze the correlation between the intensity of biomarker expression and survival of this cohort both in the observation and in the interferon-treated groups.
* To examine the prognostic role of these biomarkers on the outcome associated with melanoma in the EST-1690 cohort using quantitative-PCR.
* To isolate RNA from the primary specimens from patients enrolled in the EST-1690 cohort to assess the expression of genes suggested by cDNA microarray and IHC analyses (e.g., NCOA3, SPP1, and RGS1) as prognostic or predictive markers.

OUTLINE: Samples from the EST-1690 cohort are obtained and analyzed for several biomarkers (i.e., NCOA3, SPP1, and RGS1) via immunohistochemistry and quantitative PCR. RNA is isolated from the specimens to assess gene expression via quantitative PCR.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of melanoma

  * No metastatic disease at diagnosis
* Treated on protocol EST-1690
* Primary tumor tissue specimens available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients enrolled on E1690
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2011-02-08 (Actual); Primary Completion 2011-08-08 (Actual); Study Completion 2011-08-08 (Actual)

PRIMARY OUTCOMES:
Prognostic role of several biomarkers on the outcome associated with melanoma using IHC | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Kashani-Sabet, MD, Study Chair — University of California, San Francisco